CLINICAL TRIAL: NCT02258893
Title: Indoor Nitrogen Dioxide Exposure and Children With Asthma: An Intervention Trial
Brief Title: Indoor Air Pollution and Children With Asthma: An Intervention Trial
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Harvard University (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1308012531; 5R01ES023505-05 (NIH)
Record Dates: First submitted 2014-10-02; First posted 2014-10-08 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Nitrogen Dioxide; Parts per billion
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- NO2 Scrubber, then HEPA filter, then Control (Experimental): Participants will have 3 periods of 4 weeks with each filter with a 1 week washout between phases in the order of NO2 Scrubber, then HEPA filter, then Control.
  Interventions: Other: NO2 Scrubber; Other: HEPA filter; Other: Control
- NO2 Scrubber, then Control, then HEPA filter (Experimental): Participants will have 3 periods of 4 weeks with each filter with a 1 week washout between phases in the order of NO2 Scrubber, then Control, then HEPA filter
  Interventions: Other: NO2 Scrubber; Other: HEPA filter; Other: Control
- HEPA filter, then NO2 scrubber, then Control (Experimental): Participants will have 3 periods of 4 weeks with each filter with a 1 week washout between phases in the order of HEPA filter, then NO2 scrubber, then Control
  Interventions: Other: NO2 Scrubber; Other: HEPA filter; Other: Control
- HEPA filter, then Control, then NO2 scrubber (Experimental): Participants will have 3 periods of 4 weeks with each filter with a 1 week washout between phases in the order of HEPA filter, then Control, then NO2 scrubber
  Interventions: Other: NO2 Scrubber; Other: HEPA filter; Other: Control
- Control, then HEPA filter, then NO2 scrubber (Experimental): Participants will have 3 periods of 4 weeks with each filter with a 1 week washout between phases in the order of Control, then HEPA filter, then NO2 scrubber
  Interventions: Other: NO2 Scrubber; Other: HEPA filter; Other: Control
- Control, then NO2 scrubber, then HEPA filter (Experimental): Participants will have 3 periods of 4 weeks with each filter with a 1 week washout between phases in the order of Control, then NO2 scrubber, then HEPA filter
  Interventions: Other: NO2 Scrubber; Other: HEPA filter; Other: Control

INTERVENTIONS:
Other: NO2 Scrubber — an NO2 scrubber that removes NO2 and particles
Other: HEPA filter — a HEPA filter that removes 95% of suspended particles ≥ 0.003 μm in size (but does not remove NO2)
Other: Control — a "control" filter designed to be the same size and weight as the other two filters, but filters neither NO2 nor particles

SUMMARY:
The purpose of this study is to determine whether reducing indoor exposure to NO2 and particles improves respiratory health in children with asthma.

DETAILED DESCRIPTION:
We have designed a randomized, double-blind, triple cross-over intervention study to examine the efficacy of indoor NO2 reduction on reducing asthma severity. Since particles and NO2 are both byproducts of combustion and associated with gas stove use, the intervention protocol includes a condition using a filter designed to remove particles also implicated in asthma exacerbations (e.g., coarse, fine and ultrafine particles including airborne mold spores and allergens) while leaving NO2 virtually untouched. Primary and secondary aims of the trial include, respectively, determining whether reducing exposure to NO2 and particles compared to a "control" (non-filtered) condition results in a clinically significant reduction in asthma severity measured by a difference in days of symptoms between intervention arms.

Families with asthmatic children age 5-11 will be recruited from selected communities using a: (1) flyers distributed in elementary schools, (2) postcards send to families from purchased mailing lists, (3) posters placed in community buildings (libraries, clinics, etc.), (4) online (Facebook, Craigslist), and (5) letter mailed to families targeted through Yale Joint Data Analytics Team (JDAT). Volunteers will be screened for preliminary eligibility based on household characteristics and active asthmatic status. Potentially eligible families will have homes with a gas cooking stove and seven rooms or fewer. Potentially eligible children will be aged 5-11; have asthma symptoms and/or medication use consistent with severity score categories 2 (mild persistent), 3 (moderate), or 4 (severe) during the previous 12 months; and reside at least 5 days and nights every week in the eligible home.

Households meeting these preliminary criteria will be asked to participate in passive NO2 sampling. A single Palmes tube will be sent to the home for placement in the main living space for one week. Families will be called after one week and instructed to cap and return the NO2 monitor in a pre-paid mailer. Families of children living in homes where the one-week integrated average NO2 concentration is ≥ 15 ppb will be invited to participate. We will permit enrollment of more than one eligible child per family. Participating families will be randomized into one of 6 treatment sequences each requiring 3 periods of 4-weeks preceded by a 1-week washout period. Randomization will be blocked so that for every 18 subjects randomized there will be 3 in each sequence. Randomization will be conducted blindly by the data management department such that each scheduled initial interview/air cleaner installation is assigned a treatment sequence (referring to machines and filters already on site). Minimization techniques will be used to balance the randomized allocation as necessary. Total subject participation time up to 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 5-11 years of age, enrolled in grades K-5 and living in the recruitment area (CT, MA)
* [The screening questionnaire will determine asthma symptoms in the past 12 months (wheeze, persistent cough, shortness of breath, chest tightness); and asthma medication use in the past 12 months (short-acting β2-agonists, long-acting β2-agonists, inhaled steroids, oral steroids, theophylline, cromones, and/or leukotriene inhibitors). Based on symptoms and medication, asthma severity will be categorized with a score adapted from the Global Initiative for Asthma guidelines (1=mild transient, 2=mild persistent, 3=moderate, 4=severe). Only children in categories 2 (mild persistent, 3 (moderate) or 4 (severe) will be eligible.]
* For potential subjects satisfying these inclusion criteria, a passive NO2 monitor will be sent to the home for placement in the main living space for one week. Families will be called after one week and instructed to cap and return the NO2 monitor in a pre-paid mailer. Families of children living in homes where the one-week integrated average NO2 concentration is ≥ 15 ppb will be invited to participate. We will permit the enrollment of more than one eligible child per family.

Exclusion Criteria:

* Using steroid medication for a condition other than asthma
* Chronic respiratory condition other than asthma
* Intention to move or relocate within 6 months

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Days with symptoms | Final 14 days of intervention
  The maximum of the following variables reported over the 2-week recall period: (1) number of days with wheezing, chest tightness, or persistent cough; (2) number of nights of sleep disturbance; (3) number of days when activities were affected.

SECONDARY OUTCOMES:
Days of wheeze | Post 4 week intervention
  As measured by self report
Night symptoms | Post 4 week intervention
  As measured by self report
Rescue medication use | Post 4 week intervention
  As measured by self report
Symptom Score | Last 4 weeks of intervention
  The score is adapted from the Global Initiative for Asthma Guidelines which incorporates type and frequency of symptoms and medications. The symptom score portion, is a 5-level score calculated based on symptoms during the last 4-weeks of the intervention.
Amount of Restricted Activity | Post 4 week intervention
  Activity Restrictions as measured by self report
Number of Missed days of school | Post 4 week intervention
  As measured by self report
Number of Hospitalizations | Post 4 week intervention
  As measured by self report
Number of Emergency Room Visits | Post 4 week intervention
  As measured by self report
Number of Doctors Visits | Post 4 week intervention
  As measured by self report

CONTACTS AND LOCATIONS:
Overall Officials: Brian Leaderer, PhD, MPH, Principal Investigator — Yale University; Michael Bracken, PhD MPH FACE, Principal Investigator — Yale University; Theodore Holford, PhD, Principal Investigator — Yale University; Janneane Gent, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Gent JF, Holford TR, Bracken MB, Plano JM, McKay LA, Sorrentino KM, Koutrakis P, Leaderer BP. Childhood asthma and household exposures to nitrogen dioxide and fine particles: a triple-crossover randomized intervention trial. J Asthma. 2023 Apr;60(4):744-753. doi: 10.1080/02770903.2022.2093219. Epub 2022 Jul 7. PMID 35796019